CLINICAL TRIAL: NCT00407524
Title: AKL1 Asthma Study - Randomised, Double-Blind, Placebo Controlled, Cross Over Study to Determine Safety and Efficacy of Oral AKL1 in Treating Patients With Asthma
Brief Title: AKL 1 Asthma Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 03GP013
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: AKL 1

SUMMARY:
This study aims to provide scientific evidence of the efficacy and safety of this agent as 'add-on' therapy for adult patients whose asthma remains uncontrolled on standard medication. The aims are to assess the efficacy, safety and tolerability of AKL 1 companred to placebo in the treatment of asthma.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is of either sex and between the ages of 18 to 70 years, inclusive.
2. The patient has received verbal and written study information, all questions have been answered satisfactorily and a consent form has been personally signed and dated by the patient and the investigator.
3. The patient has a diagnosis of persistent chronic bronchial asthma (with reference to the Global Initiative for Asthma (GINA) guidelines, NIH, NHLBI. Global Initiative for asthma. NIH Publication no.96-3659B. Bethesda, MD:NID 1998) ).
4. The patient has a FEV1 (% predicted) of > 60% at Visit 1.
5. The patient has a positive reversibility test (or history of such) with >or equal 15% improvement in FEV1 from 15 to 30 minutes after inhalation of at least 200 ug of salbutamol (beta-2-adrenergic agonist administration) or PEF variability of 20% as described in current BTS/SIGN guidelines (British Thoracic Society, Scottish Intercollegiate Guideline Network. British Guidelines on the Management of Asthma. Thorax 2003;58:1-94.
6. Females must be postmenopausal (> 1 year), surgically sterile or using adequate contraception (hormonal contraception, intrauterine device), not breast-feeding and have a negative serum pregnancy test.
7. The patient is in satisfactory health with the exception of asthma as determined by the investigator on the basis of medical history and physical examination.
8. In the investigator's judgment, the patient is able and willing to comply with Study Visits and procedures (including laboratory tests, lung function tests), and accurate and timely completion of an electronic asthma diary

Exclusion Criteria:

1. The patient has poorly controlled asthma defined as requiring a course of oral or parenteral corticosteroids, admission to hospital for asthma (including treatment in an emergency room), or exacerbation of asthma in the three months prior to Visit 1 (in the investigator's judgment).
2. Maintenance oral corticosteroid treatment.
3. The patient has seasonal asthma alone.
4. Use of unlicensed doses of inhaled corticosteroid medication (>2000mcg beclomethasone diproprionate/ day or equivalent).
5. The patient has any known laboratory abnormality, which in the opinion of the investigator, would contraindicate study participation, including, blood urea nitrogen (BUN), aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >or equal 1.5 x upper limit of normal (ULN) or creatinine > 1.5 mg/dL.
6. The patient is unable to discontinue short-acting beta-2-adrenergic agonists for at least 4 hours prior to the Screening Visit.
7. The patient has chronic heart failure class III or IV (New York Heart Association).
8. The patient has a recent (less than six months) history of stroke, transient ischemic attack or myocardial infarction.
9. The patient has a history of known alcohol or substance abuse within the one-year prior to Visit 1.
10. The patient is not able to follow study procedures (e.g., language problems, psychological disorders) or is considered to be non-compliant according to the investigator.
11. The patient has an active malignancy of any type or history of a malignancy (with the exception of patients with malignancy surgically removed with no evidence of recurrence within five years before enrolment, and patients with history of treated basal cell carcinoma).
12. The patient has any other severe or acute or chronic medical or psychiatric conditions that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
13. The patient has significant uncontrolled chronic disease, such as hepatic or renal insufficiency, which in the opinion of the investigator, would contraindicate study participation or confound interpretation of the results.
14. The patient has difficulty swallowing capsules or tablets, dysphagia or is unable to tolerate oral medication.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-10; Study Completion 2005-03

PRIMARY OUTCOMES:
mean improvements in morning prebronchodilator peak expiratory flow rate in the final week of twelve week active treatment
improvement in forced expiratory volume in one second FEV one following twelve weeks of active treatment
evaluation of adverse events
vital signs
clinial laboratory results including tests of liver function

CONTACTS AND LOCATIONS:
Overall Officials: Mike Thomas, Principal Investigator — University of Aberdeen
Locations (1):
- ACCRU, Aberdeen, United Kingdom